CLINICAL TRIAL: NCT00663611
Title: Growth Hormone Administration and the Human Immune System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999907260; 07-AG-N260; NCT00663676 (obsolete NCT alias)
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-06-06

CONDITIONS: Healthy Volunteers
Keywords: Immune Function; Metabolism; Pulsatile Growth Hormone
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study I and IB (Experimental): Each involve six subjects and are designed to test the hypothesis that pulsatile subcutaneous infusion of GH via a subcutaneous infusion pump will yield a reasonable pulsatile GH pattern. The dose of GH used in Study IB will be three-fold higher than that in Study I. Study I and IB will be done first before proceeding to Study II
  Interventions: Drug: Norditropin
- Study II (Experimental): Is a randomized, double-blinded, placebo-controlled 12 week study involving 26 subjects divided into 2 groups: Group A and Group B. Group A will involve 13 subjects receiving pulsatile GH or placebo infusion for 4 weeks with 8 week washout after intervention. Group B will involve 13 subjects receiving conventional once a day subcutaneous infusion of GH or placebo for 4 weeks with 8 week washout after intervention.
  Interventions: Drug: Norditropin; Drug: Placebo

INTERVENTIONS:
Drug: Norditropin — Norditropin (somatropin, rDNA origin) is a polypeptide hormone of recombinant DNA origin. The amino acid sequence of the product is identical to that of the human growth hormone of pituitary origin.
Drug: Placebo — 0.9% normal saline
  Arms: Study II

SUMMARY:
Background:

- In elderly individuals, an age-associated decline in the immune system s ability to function is believed to contribute to increased incidence of infection, autoimmune disorders, and cancer. This decline in immune system function may be related to the decline in the body s production of growth hormone, which helps regulate human development and may contribute to the health of the immune system. Researchers are interested in studying whether growth hormone, given as an infusion over time, can improve the function of the immune system and other body systems associated with good health.

Objectives:

- To study the effects of growth hormone administration on the immune systems of healthy men.

Eligibility:

- Healthy men between 25 and 50 years of age.

Design:

* This protocol will involve three separate studies: Study I, Study IB, and Study II. Participants in Study I and Study IB may participate in Study II as directed by the researchers.
* Participants will be screened with a full medical history and physical examination, and will provide blood, urine, and stool samples; have a glucose tolerance test; and have other tests as required by the researchers.
* Participants will have an infusion pump with a small catheter inserted beneath the skin to administer the study chemicals (either growth hormone or placebo).
* Study I and Study IB participants will receive pulses of growth hormone through the infusion pump at regular intervals to monitor the body s response to the hormone. Study IB participants will receive a higher dose of growth hormone than Study I participants.
* Throughout the study period, all participants will have frequent blood and urine tests, as well as tests of glucose tolerance and metabolism, imaging studies, and other tests as required by the researchers.
* Study II participants will be divided into two groups. The first group will receive pulses of either growth hormone or placebo infusion at intervals throughout the day for 4 weeks, followed by an 8-week period without infusions. The second group will receive conventional once-a-day infusion of growth hormone or placebo for 4 weeks, followed by an 8-week period without infusions.
* Throughout the study period, all participants will have frequent blood and urine tests, as well as tests of glucose tolerance and metabolism, imaging studies, and other tests as required by the researchers.

DETAILED DESCRIPTION:
Objectives and Specific Aims:

We plan to investigate whether growth hormone, administered in a physiological or pulsatile fashion, can elicit relevant changes in the human immune system while at the same time associated with no change or even an improvement in the metabolic profiles such as insulin sensitivity.

Experimental Design and Methods:

Thirty-eight healthy men, age 25-50, will be recruited for this study. There are three parts to this study: Study I, Study IB and Study II. Study I and IB each involve six subjects and are designed to test the hypothesis that pulsatile subcutaneous infusion of GH via a subcutaneous infusion pump yields a reasonable pulsatile GH pattern. The dose of GH used in Study IB is three-fold higher than in Study I. Study I and IB are done first before proceeding to Study II.

Study II is a randomized, double-blinded, placebo-controlled 12-week study involving 26 subjects divided into 2 groups: Group A and Group B. Group A involves 13 subjects receiving pulsatile GH or placebo infusion for 4 weeks with 8-week washout after intervention. Group B involves 13 subjects receiving conventional once a day subcutaneous infusion of GH or placebo for 4 weeks with 8-week washout after intervention.

Medical Relevance and Expected Outcome:

This study ascertains the significance of the effect of pulsatile growth hormone administration on the human immune system and metabolic profile.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy men only (There is a gender difference in GH response with adult females requiring on average twice the GH dose for similar effects. In order to eliminate gender difference as a confounding factor in this study, we are studying male subjects only because the GH dose requirement is lower.)
  2. Age 25-50 (Age restriction is used to remove age as a confounding factor because GH and thymic function are known to decrease with age.)
  3. Screening laboratory evaluations with no clinically significant abnormal results (minor deviations from "normal" lab results will be at the discretion of the principal investigator):

     1. fasting comprehensive metabolic panel
     2. complete blood count with differential and platelets
     3. 75-gram oral glucose tolerance test (OGTT)

        * fasting plasma glucose (FPG) < 100 mg/dL
        * 2-hr OGTT < 140 mg/dL
     4. Insulin-like growth factor-I (IGF-I)
     5. thyroid function test (TSH, free T3, free T4)
     6. fasting lipid profile
  4. BMI < 30 (Men with BMI >= 30 are excluded because decrease in GH secretion and clearance has been shown in obesity.)
  5. Have NOT participated in another clinical trial involving any pharmacologic agents within the past 60 days
  6. Able to complete an inform consent
  7. Agree to not participate in other clinical trials within the study period

EXCLUSION CRITERIA:

1. Women
2. FPG >= 100 mg/dL or 2-hour OGTT >= 140 mg/dL
3. Abnormal electrocardiogram (EKG) suggesting possible underlying cardiac conditions that, in the opinion of the investigator(s), may cause participation of the subject in the study unsafe
4. Positive stool guaiac
5. Evidence of illicit drug use
6. History of smoking any tobacco products within one year prior to screening
7. Alcohol intake > 30 grams (drink more than 2 beers per day OR equivalent amount of alcohol)
8. History of Human Immunodeficiency Virus (HIV) infection
9. History of active or chronic Hepatitis B and/or C infection
10. History of malignancy
11. History of coronary disease
12. History of seizures or other neurologic diseases
13. History of liver or renal diseases
14. History of gastrointestinal or endocrine disorders
15. History of glucocorticoid use (over one month) or other immunosuppressive agents (any)
16. unable to undergo a magnetic resonance imaging (MRI) procedure
17. Any medical history that, in the opinion of the investigator(s), will make participation of the subject in the study unsafe

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2006-10-19; Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-06 (Actual)

PRIMARY OUTCOMES:
GH administration may elicit clinical significant and relevant changes in the human immune system | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chee W Chia, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.

REFERENCES:
- [Background] Bar-Dayan Y, Small M. Effect of bovine growth hormone administration on the pattern of thymic involution in mice. Thymus. 1994;23(2):95-101. PMID 7725388
- [Background] Napolitano LA, Lo JC, Gotway MB, Mulligan K, Barbour JD, Schmidt D, Grant RM, Halvorsen RA, Schambelan M, McCune JM. Increased thymic mass and circulating naive CD4 T cells in HIV-1-infected adults treated with growth hormone. AIDS. 2002 May 24;16(8):1103-11. doi: 10.1097/00002030-200205240-00003. PMID 12004268
- [Background] Murphy WJ, Durum SK, Longo DL. Role of neuroendocrine hormones in murine T cell development. Growth hormone exerts thymopoietic effects in vivo. J Immunol. 1992 Dec 15;149(12):3851-7. PMID 1460277